CLINICAL TRIAL: NCT05175352
Title: A Phase 1, Open-label, Single-sequence Study to Evaluate Potential Disease-mediated Drug-drug Interaction With Selected Cytochrome P450 Substrates in Adult Subjects With Active Eosinophilic Esophagitis Receiving Cendakimab
Brief Title: A Study Evaluating Potential Disease-Mediated Drug-Drug Interaction in Adult Participants With Active Eosinophilic Esophagitis Receiving Cendakimab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-93538-DDI-001
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Cendakimab; Drug-drug interactions; DDI
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — cendakimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of Cendakimab and Cytochrome P450 (CYP) substrates (Experimental)
  Interventions: Drug: Cendakimab; Drug: CYP substrates

INTERVENTIONS:
Drug: Cendakimab — Specified dose on specified days
  Other Names: CC-93538; BMS-986355
Drug: CYP substrates — Specified dose on specified days

SUMMARY:
The purpose of this study to evaluate the potential for disease-mediated drug-drug interactions between cendakimab and selected substrates of metabolic enzymes in eosinophilic esophagitis participants.

ELIGIBILITY:
Inclusion Criteria:

* Active Eosinophilic esophagitis (EoE) with histologic evidence as a peak count of ≥ 15 eosinophils per higher-power field at any 2 levels of the esophagus
* Previously received an adequate trial of proton-pump inhibitor medication that did not provide complete response to EoE
* EoE symptoms documented in daily diary during the screening period

Exclusion Criteria:

* On a regimen of therapeutic anticoagulation
* Demonstrates evidence of immunosuppression or is receiving systemic immunosuppressive or immunomodulating drugs
* Currently receiving a high potency topical corticosteroid for dermatologic use

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Area under the concentration-time curve calculated from time zero to infinity (AUC0-∞) | Up to 18 Weeks
Pharmacokinetics - Area under the concentration-time curve calculated from time zero to 12 hours postdose (AUC0-12h) | Up to 18 Weeks

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum plasma concentration of drug (Cmax) | Up to 18 Weeks
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to 34 Weeks
Severity of TEAEs | Up to 34 Weeks
Relationship of TEAEs | Up to 34 Weeks
Immunogenicity profile of cendakimab measured by assessment of the presence of specific anti-drug antibodies (ADAs) over time | Up to 34 Weeks
Number of participants with clinical laboratory abnormalities | Up to 34 weeks
Number of participants with electrocardiogram abnormalities | Up to 34 weeks
Number of participants with vital sign abnormalities | Up to 34 weeks
Number of participants with physical examination sign abnormalities | Up to 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (12):
  - Local Institution - 004, Tucson, Arizona
  - Local Institution - 001, Los Angeles, California
  - Local Institution - 022, San Diego, California
  - Local Institution - 016, Bristol, Connecticut
  - Local Institution - 002, Inverness, Florida
  - Local Institution - 010, Miami, Florida
  - Local Institution - 021, Plantation, Florida
  - Local Institution - 020, Gurnee, Illinois
  - Local Institution - 008, Iowa City, Iowa
  - Local Institution - 003, Albuquerque, New Mexico
  - Local Institution - 018, Durham, North Carolina
  - Local Institution - 012, Columbus, Ohio

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com